CLINICAL TRIAL: NCT05912309
Title: Effects of Time-restricted Eating and Exercise Training on Skeletal Muscle Mass Quantity, Quality and Function in Postmenopausal Women With Overweight and Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Idoia Labayen (Other)
Collaborators: Hospital of Navarra (Other)
Responsible Party: Sponsor-Investigator, Idoia Labayen, Senior Lecturer, Universidad Pública de Navarra
Organization: Universidad Pública de Navarra (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI_2023/8; EXP_75091 (Other Grant/Funding Number: Centro Superior de Deportes (CSD))
Record Dates: First submitted 2023-05-17; First posted 2023-06-22 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Menopause Related Conditions; Sarcopenia; Osteoporosis Postmenopausal; Obesity
Keywords: Obesity; Overweight; Sarcopenia; Menopause; Exercise; Resistance Exercise; Physical activity; intramuscular adipose tissue; Visceral adipose tissue; Liver fat; Skeletal muscle mass; Muscle function; Muscle quality; Osteoporosis
MeSH Terms: conditions — Sarcopenia; Osteoporosis, Postmenopausal; Obesity; Overweight; Motor Activity; Fatty Liver; Osteoporosis | interventions — Exercise; Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel-arm clinical trial
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time Restricted Eating (TRE) (Experimental)
  Interventions: Behavioral: Time Restricted Eating (TRE)
- Time Restricted Eating (TRE) + Exercise (Experimental)
  Interventions: Behavioral: Time Restricted Eating (TRE); Behavioral: Exercise
- Caloric restriction (CR) + Exercise (Active Comparator)
  Interventions: Behavioral: Exercise; Behavioral: Caloric Restriction

INTERVENTIONS:
Behavioral: Time Restricted Eating (TRE) — Participants will be required to reduce their eating time window to ≤ 8 hours/day. Women can choose when to begin eating, but the last meal should be completed before or at 20:00 hours (concentrating the eating window towards the active phase confers higher cardiometabolic health benefits). Our preliminary results suggest that this eating window is feasible and safe. Participants will receive dietary advice regarding the daily amount of high quality protein and meal-specific protein quantities. All the participants will attend a lifestyle education program based on Mediterranean diet and WHO physical activity recommendations every two weeks.
  Arms: Time Restricted Eating (TRE); Time Restricted Eating (TRE) + Exercise
Behavioral: Exercise — Sport sciences specialists will design, supervise and monitor the concurrent exercise intervention following the 2020 WHO recommendations. The program will be tailored to the participant's ability and health, and will be focused on a gradual increase to levels that are safe. Resistance training: 3 times/week designed to manage, attenuate and even prevent the loss of skeletal muscle tissue and function. The exercise sessions will be scheduled within or immediately after their eating window in order to maximize muscular muscle protein synthesis. Morning and afternoon training schedules will be offered to participants.
  Arms: Caloric restriction (CR) + Exercise; Time Restricted Eating (TRE) + Exercise
Behavioral: Caloric Restriction — Individualised intensive behavioural intervention weight loss program including CR, exercise training and lifestyle education designed according to the current guidelines. CR will be tailored to participants (objectively assessed). Diet will provide 600 kcal/day less than the individual energy requirements based on measured resting energy expenditure (indirect calorimetry) and multiplied by an activity factor obtained by accelerometry. Experienced nutritionists will design personalized and balanced CR diet, and will train the participants through the food exchange system to follow the treatment. In those cases in which the CR compromised a protein intake of at least 1.2 g/kg/day, the macronutrient percentage distribution will be modified prioritizing achieving this minimum protein intake.
  Arms: Caloric restriction (CR) + Exercise

SUMMARY:
The goal of this randomized controlled trial] is to investigate the effects of a 12-week time restricted eating (TRE) and exercise combined intervention, as compared to (i) TRE alone, and to (ii) Caloric Restriction (CR) plus the same exercise intervention elicited by the TRE group, on Skeletal muscle tissue (SMT) quantity, quality and function (primary outcome), Resting energy expenditure (REE) and cardiometabolic health (secondary outcomes), and miRNA biomarkers in postmenopausal women with overweight or obesity.

DETAILED DESCRIPTION:
Time restricted eating (TRE) may be a potential lifestyle tool for the management of obesity in populations at risk of sarcopenia. However, weight loss may occur at the expense of lean mass, thus producing an undesirable reduction of Skeletal Muscle Tissue (SMT). To date, studies focused on body composition suffer from methodological shortcomings in adequate SMT quantity and quality measurement (e.g. using gold standard magnetic resonance imaging, MRI) and function, dietary intake protein counselling and the monitoring of dietary energy and macronutrient intake. Importantly, no TRE studies have been conducted in postmenopausal women with overweight who are at high risk of sarcopenia. Studies such as the one presented herein are needed to elucidate the effects of TRE on SMT and protein balance in the middle- and long-term lifestyle intervention. In addition, the potentially myoprotective roles of dietary protein and exercise need to be more cogently established within the framework of a TRE regime in populations at risk of sarcopenia. Further, the effects of TRE+exercise on SMT quantity, quality and function should be compared to currently accepted lifestyle therapy lifestyle therapy for obesity management in adults at high risk of sarcopenia (Caloric Restriction (CR) + exercise and adequate protein intake). Finally, the underlying mechanisms of SMT quantity, quality and function loss, as well as those explaining the effects of TRE and exercise are unknown. The investigators will explore circulating miRNA profiles as novel, non-invasive and feasible prognostic biomarkers of changes in SMT quantity, quality and function.

* This study will be the first randomized controlled trial to investigate whether the addition of exercise to TRE is able to reverse the SMT loss induced by the TRE alone, and if the combination of TRE and exercise confers any additional benefits on SMT quantity, quality and function above the currently recommended lifestyle intervention.
* The few previous TRE studies examined changes in body composition using dual-energy X-ray absorptiometry (DXA); however, this is not the most appropriate method to assess SMT and it does not evaluate IMAT. The investigators will use magnetic resonance imaging (MRI) scanning (gold standard) to measure changes in SMT and intra-muscular adipose tissue (IMAT, muscle quality).
* There is a lack of knowledge on the effects of TRE on muscle strength. This important determinant of sarcopenia will be assessed with gold standard methodology.
* This study will be pioneer at quantifying the long-term adherence and the persistence of the effects of TRE and exercise on SMT quantity, IMAT and function (12 months)
* Importantly, the investigators will be able to study miRNA predictors of changes in SMT quantity, IMAT and function in postmenopausal women.
* Available studies on TRE, although enlightening, have solely assessed acute or short-term (<2 weeks) effects of TRE on Resting Energy Expenditure (REE). It will be evaluated whether TRE and exercise confers any additional advantage on REE maintenance above the currently recommended lifestyle intervention in the middle and long-term.
* The majority of TRE studies were focused on body weight or total adiposity. The present study will also evaluate the effects of the intervention on specific ectopic fat depots strongly associated with cardiometabolic health, morbidity and mortality using MRI (i.e., visceral adipose tissue (VAT) and liver fat), in the middle- (12 weeks) and long-term (12 months).
* Impaired systemic glucose homeostasis is common in postmenopausal women with overweight. TRE and exercise intervention has the potential of reducing Insulin Resistance (IR); therefore, the present project will include the measurement of continuous glucose monitoring (CGM) analyzing day-to-day glucose homeostasis.
* Exercise reduces the risk of sarcopenic obesity and ectopic fat aggregation, improves cardiometabolic health and reduces proinflammatory markers, but the underlying mechanisms are largely unknown. The analysis of circulating miRNA profiles can help to elucidate the mechanisms explaining the response to the lifestyle intervention as well as identifying potential therapeutic targets.
* There is a high inter-individual variability in the response to TRE and exercise interventions, but its predictors are unknown. This study will focus on miRNAs as potential predictive and prognostic biomarkers.
* Gender dimension: women are under-represented in TRE studies and there is no previous study conducted on postmenopausal women. Studies on this specific population are of great interest for several reasons: unique hormonal status that confers elevated risk of obesity and obesity-related morbidities, high risk of sarcopenia, and an enormous interest on self-administered TRE that could entail unknown health consequences.

Participants: Postmenopausal women (n=78) with an absence of menses for over two years (at least stage +1a) and with overweight (BMI>25 kg/m2) or obesity (BMI>30 kg/m2 and BMI<=40 kg/m2) will be recruited at the Endocrinology Unit of the University Hospital of Navarra.

Intervention: Participants will be randomly allocated 1:1:1 to (1) CR+exercise, (2) TRE, and (3) TRE+exercise groups. Before baseline measurements and group allocation, there will be a 2-week lead-in period where the eating window, glucose and physical activity will be continuously monitored. Thereafter, participants will follow the 12-week intervention according to their allocated group.

* CR+exercise group: Individualized intensive behavioral intervention weight loss program including CR, exercise training and lifestyle education designed according to the current guidelines. CR will be tailored to participants (objectively assessed). Diet will provide 600 kcal/day less than the individual energy requirements based on measured REE (indirect calorimetry) and multiplied by an activity factor obtained by accelerometry. Experienced nutritionists will design personalized and balanced CR diet, and will train the participants through the food exchange system to follow the treatment. In those cases in which the CR compromised a protein intake of at least 1.2 g/kg/day, the macronutrient percentage distribution will be modified prioritizing achieving this minimum protein intake. Sport sciences specialist will design, supervise and monitor the concurrent exercise intervention following the 2020 WHO recommendations. The program will be tailored to the participant ́s ability and health, and will be focused on a gradual increase to levels that are safe. Resistance training: 2-3 times/week designed to manage, attenuate and even prevent the loss of SMT and function.
* TRE group: Participants will be required to reduce their eating time window to ≤ 8 hours/day. Women can choose when to begin eating, but the last meal should be completed before or at 20:00 hours (concentrating the eating window towards the active phase confers higher cardiometabolic health benefits). Our preliminary results suggest that this eating window is feasible and safe.
* TRE+exercise group: This group will combine the intervention of the TRE group and the same exercise intervention of the CR+exercise group. The exercise sessions will be scheduled within or immediately after their eating window in order to maximize MPS. Morning and afternoon training schedules will be offered to participants.

The three groups will receive dietary advice regarding the daily amount of high quality protein and meal-specific protein quantities. All the participants will attend a lifestyle education program based on Mediterranean diet and WHO physical activity recommendations every two weeks.

Long-term follow-up: Weight cycling is frequent in women and is associated with increased morbidity. There are no previous studies examining the persistence of the effects of TRE+exercise in the long-term. Also, it seems that the adherence to the TRE regime is higher than to the CR, but the evidence is scarce. This project will assess the main study outcomes and the adherence in order to examine the persistence and feasibility of the intervention effects 12 months after the cessation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 65 years.
* Menopause (Phase +1a)
* Body mass index ≥25.0 and <40 kg/m2 or waist circumference > 94 cm.
* Weight stability (within 3% of screening weight) for >3 months prior to baseline.
* Sedentary lifestyle (<150 min/week of moderate-vigorous intensity exercise) for >3 months prior to baseline.
* Usual feeding window ≥12 hours.

Exclusion Criteria:

* History of major adverse cardiovascular events, clinically significant renal, endocrine or neurological disease, bariatric surgery, HIV/AIDS, known inflammatory and/or rheumatologic disease, cancer or other medical condition in which fasting or exercise is contraindicated.
* Use of exogenous (sex) hormones (hormone replacement therapy).
* Type 1 or type 2 diabetes.
* Severe psychiatric disorders, eating disorders, sleep disorders or alcohol abuse.
* Regular use of medications or compounds that may affect study results.
* Participating in a weight loss or weight control program.
* Caregiver of a dependent person who requires frequent nighttime care/sleep interruptions. Shift workers with variable schedules (e.g., nighttime). Frequent travel across time zones during the study period.
* Fear of needles and claustrophobia of magnetic resonance imaging (MRI).
* Any medical situation that prevents the performance of MRI (pacemakers, prostheses, etc).
* Being unable to understand and accept the instructions or the objectives and protocol of the study.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle tissue quantity - Baseline | Just after the end of the 12-week intervention (+1 to +3 days)
  Skeletal muscle tissue (Cross sectional area (cm2) and Volume (cm3)) will be quantified by magnetic resonance imaging ((MRI) Magnetom Vida 3T system, Siemens, Healthineers), the gold standard methodology, at the most representative sites: mid-thigh, psoas (L3) and paraspinal and abdominal wall (L2-L4). Both Detailed information about imaging segmentation and processing can be found in previous work of our group. The segmentation for all these structures will be done with a semiautomatic proprietary algorithm developed in our group.
Skeletal muscle tissue quantity - 12 weeks | Just before the start of the 12-week intervention (-3 to -1 days), just after the end of the 12-week intervention (+1 to +3 days) and 1 year after the end of the intervention
  Skeletal muscle tissue (Cross sectional area (cm2) and Volume (cm3)) will be quantified by magnetic resonance imaging ((MRI) Magnetom Vida 3T system, Siemens, Healthineers), the gold standard methodology, at the most representative sites: mid-thigh, psoas (L3) and paraspinal and abdominal wall (L2-L4). Both Detailed information about imaging segmentation and processing can be found in previous work of our group. The segmentation for all these structures will be done with a semiautomatic proprietary algorithm developed in our group.
Skeletal muscle tissue quantity - 1 year | 1 year after the end of the intervention
  Skeletal muscle tissue (Cross sectional area (cm2) and Volume (cm3)) will be quantified by magnetic resonance imaging ((MRI) Magnetom Vida 3T system, Siemens, Healthineers), the gold standard methodology, at the most representative sites: mid-thigh, psoas (L3) and paraspinal and abdominal wall (L2-L4). Both Detailed information about imaging segmentation and processing can be found in previous work of our group. The segmentation for all these structures will be done with a semiautomatic proprietary algorithm developed in our group.
Skeletal muscle tissue quality - Baseline | Just before the start of the 12-week intervention (-3 to -1 days)
  Intermuscular and Intramuscular adipose tissue (fat fraction(%)) will be quantified by magnetic resonance imaging ((MRI) Magnetom Vida 3T system, Siemens, Healthineers), the gold standard methodology, at the most representative sites: mid-thigh, psoas (L3) and paraspinal and abdominal wall (L2-L4). Both Detailed information about imaging segmentation and processing can be found in previous work of our group. The segmentation for all these structures will be done with a semiautomatic proprietary algorithm developed in our group.
Skeletal muscle tissue quality - 12 weeks | Just after the end of the 12-week intervention (+1 to +3 days)
  Intermuscular and Intramuscular adipose tissue (fat fraction(%)) will be quantified by magnetic resonance imaging ((MRI) Magnetom Vida 3T system, Siemens, Healthineers), the gold standard methodology, at the most representative sites: mid-thigh, psoas (L3) and paraspinal and abdominal wall (L2-L4). Both Detailed information about imaging segmentation and processing can be found in previous work of our group. The segmentation for all these structures will be done with a semiautomatic proprietary algorithm developed in our group.
Skeletal muscle tissue quality - 1 Year | 1 year after the end of the intervention
  Intermuscular and Intramuscular adipose tissue (fat fraction(%)) will be quantified by magnetic resonance imaging ((MRI) Magnetom Vida 3T system, Siemens, Healthineers), the gold standard methodology, at the most representative sites: mid-thigh, psoas (L3) and paraspinal and abdominal wall (L2-L4). Both Detailed information about imaging segmentation and processing can be found in previous work of our group. The segmentation for all these structures will be done with a semiautomatic proprietary algorithm developed in our group.
Lower Body Muscle function - Baseline | Just before the start of the 12-week intervention (-3 to -1 days)
  Muscle function will be determined using a linear position transducer (watios and m/s). 1-RM will be also estimated from this data.
Lower Body Muscle function - 12 weeks | Just after the end of the 12-week intervention (+1 to +3 days)
  Muscle function will be determined using a linear position transducer (watios and m/s). 1-RM will be also estimated from this data.
Lower Body Muscle function - 1 year | 1 year after the end of the intervention
  Muscle function will be determined using a linear position transducer (watios and m/s). 1-RM will be also estimated from this data.
Upper Body Muscle function - Baseline | Just before the start of the 12-week intervention (-3 to -1 days)
  Muscle function will be determined using a linear position transducer (watios and m/s). 1-RM will be also estimated from this data.
Upper Body Muscle function - 12 weeks | Just after the end of the 12-week intervention (+1 to +3 days)
  Muscle function will be determined using a linear position transducer (watios and m/s). 1-RM will be also estimated from this data.
Upper Body Muscle function - 1 year | 1 year after the end of the intervention
  Muscle function will be determined using a linear position transducer (watios and m/s). 1-RM will be also estimated from this data.
Handgrip Strength - Baseline | Just before the start of the 12-week intervention (-3 to -1 days)
  Handgrip strength will be determined by the handgrip strength test using a digital hand dynamometer (kilograms)
Handgrip Strength - 12 weeks | Just after the end of the 12-week intervention (+1 to +3 days)
  Handgrip strength will be determined by the handgrip strength test using a digital hand dynamometer (kilograms)
Handgrip Strength - 1 year | 1 year after the end of the intervention
  Handgrip strength will be determined by the handgrip strength test using a digital hand dynamometer (kilograms)

SECONDARY OUTCOMES:
Resting energy expenditure | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  We will measure gas exchange to objectively determine REE and substrate oxidation rates using indirect calorimetry (Q-NRG, COSMED, Rome, Italy), the gold standard methodology, following standard procedures.
Ectopic fat | Just before the start of the 12-week intervention (-3 to -1 days), just after the end of the 12-week intervention (+1 to +3 days) and 1 year after the end of the intervention
  Visceral adipose tissue and liver fat will be also measured by MRI (Magnetom Vida 3T system, Siemens, Healthineers), the gold standard methodology as previously described.
Bone Mineral Density | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  Bone mineral density (g/cm2) will be measured by DXA (gold standard).
Lean Mass | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  Lean mass (kg) will be measured by DXA (gold standard).
Bone Mineral Content | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  Bone mineral content (g) will be measured by DXA (gold standard).
Whole body fat percentage | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  Whole body fat percentage (%) will be measured by air displacement plethysmography (BodPod, COSMED, Rome, Italy) (gold standard).
Glucose homeostasis | Just before the start of the 12-week intervention (-12 to -3 days), just after the end of the 12-week intervention (+3 to +12 days) and 1 year after the end of the intervention
  Glucose homeostasis will be evaluated with the continuous glucose monitoring over consecutive 24h/10 days.
Whole body Insulin Resistance | Just before the start of the 12-week intervention (-12 to -3 days), just after the end of the 12-week intervention (+3 to +12 days) and 1 year after the end of the intervention
  Whole body IR with the standard 75-grams two-hour oral glucose tolerance test.
Serum glucose | Just before the start of the 12-week intervention (-12 to -3 days), just after the end of the 12-week intervention (+3 to +12 days) and 1 year after the end of the intervention
  Fasting serum samples will be used to measure glucose (mg/dl)
Serum Insulin | Just before the start of the 12-week intervention (-12 to -3 days), just after the end of the 12-week intervention (+3 to +12 days) and 1 year after the end of the intervention
  Fasting serum samples will be used to measure insulin (mg/dl)
Serum adiponectin | Just before the start of the 12-week intervention (-12 to -3 days), just after the end of the 12-week intervention (+3 to +12 days) and 1 year after the end of the intervention
  Fasting serum samples will be used to measure adiponectin (μg/ml)
HOMA-IR | Just before the start of the 12-week intervention (-12 to -3 days), just after the end of the 12-week intervention (+3 to +12 days) and 1 year after the end of the intervention
  HOMA-IR will be calculated using the following formula: [fasting serum insulin (μU/mL) × Fasting serum glucose (mg/dL)/405]
Circulating total cholesterol | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  Circulating total cholesterol (mg/dL) will be measured in plasma after an overnight fast.
LDL-Cholesterol | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  LDL-Cholesterol (mg/dL) will be measured in plasma after an overnight fast.
HDL-Cholesterol | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  HDL-Cholesterol (mg/dL) will be measured in plasma after an overnight fast.
Triglycerides | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  Triglycerides will be measured in plasma after an overnight fast.
Apolipoprotein B | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  Apolipoprotein B (mg/dl) will be measured in plasma after an overnight fast.
Apolipoprotein A | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days) and 1 year after the end of the intervention
  Apolipoprotein A (mg/dl) will be measured in plasma after an overnight fast.
Micro RNA analyses | Just before the start of the 12-week intervention (-7 to -3 days) and just after the end of the 12-week intervention (+3 to +7 days)
  Expression of circulating miRNAs will be analyzed in plasma samples, using RNAseq methodology at baseline and at the end of the intervention (12-week). Briefly, total RNA will be isolate and RNA quantity and quality will be confirmed by gel electrophoresis and spectrophotometry. RNA integrity will also be assessed by 2100 Bioanalyzer of Agilent Technologies. Specific NGS library kit will be used to generate sequencing libraries. Then, fragments of 145-160bp will be selected. Library sequencing will be done on a MiSeq instrument (Illumina Inc.) using Miseq Reagent kit V3 (Illumina Inc.), 12 libraries per sequencing run will be multiplexed. Analysis of results will be performed using MiSeqReporter (MSR) software of Illumina. Sequence alignment will be done using BWA and variant calling using GATK algorithm. Changes on miRNA expression levels will be evaluated with specific software packages (SHiMPS aligner, DESeq2, miRDeep, sRNAPipe and miRNET v2.0).

OTHER OUTCOMES:
Energy intake and macronutrient distribution | Just before the start of the 12-week intervention (-7 to -3 days), every 2 weeks during the 12-week intervention, just after the end of the 12-week intervention (+3 to +7 days), and 1 year after the end of the intervention
  24h dietary recalls will be done to gather information about daily energy intake (kcals) and macronutrient distribution (Carbohydrate %, Protein % and fat %)
Physical activity | Just before the start of the 12-week intervention (-12 to -3 days), just after the end of the 12-week intervention (+3 to +12 days) and 1 year after the end of the intervention
  Participants will be asked to wear a wrist-worn GT3X+ model accelerometer (ActiGraph, Pensacola, FL, USA) for 7 consecutive days (24 h/day).
Adherence to lifestyle intervention | Just before the start of the 12-week intervention (-7 to -3 days), every 2 weeks during the 12-week intervention, just after the end of the 12-week intervention (+3 to +7 days), and 1 year after the end of the intervention
  Adherence to the eating window in TRE groups will be monitored using a smartphone App over the whole intervention. Adherence to the CR will be evaluated every two weeks using 24-h dietary recalls. The attendance to the exercise sessions will be registered.
Eating behavior | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days), and 1 year after the end of the intervention
  Eating behavior will be assessed using the Adult Eating Behavior Questionnaire (AEBQ).
Overall health | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days), and 1 year after the end of the intervention
  Overall health will be evaluated using the EuroQol 5 dimensions 5 levels (EQ-5D-5L), Rand Short Form 36 (SF-36), an adverse events questionnaire
Chronotype | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days), and 1 year after the end of the intervention
  Chronotype will be subjectively assessed using the validated Munich Chronotype Questionnaire (MCTQ).
Sleep | Just before the start of the 12-week intervention (-7 to -3 days), just after the end of the 12-week intervention (+3 to +7 days), and 1 year after the end of the intervention
  Sleep will be subjectively assessed using the validated Pittsburgh Sleep Quality Index (PSQI) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Idoia Labayen, PhD, Principal Investigator — Universidad Pública de Navarra; Estrella Petrina, PhD, Principal Investigator — Hospital of Navarra
Locations (1):
- Universidad Pública de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No